CLINICAL TRIAL: NCT01953003
Title: A Multicenter, Randomised, Phase III Study of Vinflunine Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced Breast Cancer Previously
Brief Title: Phase III Study of Vinflunine Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L00070 IN 311 B0
Record Dates: First submitted 2013-08-13; First posted 2013-09-30 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-01

CONDITIONS: Malignant Neoplasm of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — vinflunine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A : iv vinflunine plus Capecitabine (Experimental): Vinflunine dose 280 mg/m² on day 1 of each cycle every 3 weeks, Capecitabine 825 mg/m² twice daily orally for 14 consecutive days beginning on day 1 of each cycle followed by 1 week of rest.
  Interventions: Drug: vinflunine; Drug: Capecitabine
- capecitabineArm B : capecitabine (Active Comparator): 1250 mg/m² twice daily orally for 14 consecutive days beginning on day 1 of each cycle followed by 1 week of rest
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: vinflunine — intravenous administration day 1 once every 3 weeks, 280 mg/m²
  Other Names: Javlor
  Arms: Arm A : iv vinflunine plus Capecitabine
Drug: Capecitabine — Arm A : 1650 mg/m² Arm B : 2500 mg/m²
  Other Names: xeloda; from day 1 to day 14

SUMMARY:
Options for the treatment of patients who have progressed after an anthracycline and a taxane are limited. Capecitabine currently has a role in this setting, yet as many as 80% of patients do not respond to this treatment and those who respond eventually develop clinical resistance.

The antitumour activity of vinflunine has been demonstrated in patients with breast cancer after exposure to anthracycline and to taxane.

Vinflunine plus capecitabine has been shown to be a feasible combination for patients previously treated with an anthracycline and a taxane. Each drug in combination can be administered at efficacious doses.

This population has few therapeutic options with established clinical benefit. The development of a new regimen and potential new standard of care for this group is important.

* Primary objective:

  • to compare in patients with advanced breast cancer pretreated with anthracycline and taxane the efficacy of the combination of vinflunine and capecitabine with capecitabine alone, in terms of progression-free survival.
* Secondary objectives:

  * to evaluate the response rate, the time to response and the duration of response in both arms
  * to compare the disease control rate between arms
  * to evaluate the duration of disease control in both arms
  * to evaluate the overall survival in both arms
  * to evaluate safety

Methodology This multicentre, open-label, randomised, Phase III study will enrol a total of 334 patients with advanced breast cancer who have previously been treated with an anthracycline and a taxane. Patients will be randomised in a 1:1 ratio to receive VFL plus capecitabine (Arm A) or capecitabine alone (Arm B).

DETAILED DESCRIPTION:
RECIST 1.1 will be used for tumor assessment CTC - CAE version 3.0 will be used for safety assessment

ELIGIBILITY:
INCLUSION CRITERIA:

1. Written informed consent
2. Histologically or cytologically confirmed Her-2 negative carcinoma of the breast
3. Documented locally recurrent or metastatic disease not amenable to curative surgery or radiotherapy
4. One, two or three prior chemotherapy regimens including those administered in the neoadjuvant or adjuvant setting. At least one of the regimens must have been given for the treatment of advanced disease.
5. Prior treatment must have included both an anthracycline and a taxane. minimum cumulative dose of 180 mg/m² of doxorubicin or of 300 mg/m² of epirubicin
6. Documented progression on or within 12 months of the most recent chemotherapy.
7. Prior hormone therapy is allowed
8. Prior radiation therapy is allowed to less than 30% of the bone marrow
9. LMeasurable or non measurable disease defined according to RECIST V1.1
10. Adequate recovery from recent surgery
11. Estimated life expectancy superior or equal of 12 weeks
12. KPS equal or superior to 70%
13. Age equal or superior to 21 years and < 80 years
14. ANC) equal or superior to 1.5 x 109/L, platelet count equal or superior to 100 x109/L and haemoglobin > 10 g/dL.
15. Bilirubin inferior or equal to 1.5 x upper limit of normal (ULN), AST and ALT inferior or equal to 2.5 x ULN or inferior or equal to 5 x ULN in the case of liver metastases, alkaline phosphatase inferior or equal to 5 x ULN.
16. Calculated creatinine clearance superior or equal to 50 mL/min
17. Normal ECG
18. Patients on coumadin or warfarin must be on stable doses and INR inferior or equal to 3
19. Women of childbearing potential must be using a medically accepted method of contraception. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to first treatment administration.
20. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed with the patient before registration in the trial.

EXCLUSION CRITERIA

1. Known or with clinical evidence of brain metastasis or leptomeningeal involvement.
2. Pulmonary lymphangitis or symptomatic pleural effusion (grade > 2) that results in pulmonary dysfunction requiring active treatment.
3. Patients having received any other experimental drug or chemotherapy within 30 days
4. History of second primary malignancy, except: bilateral breast carcinoma, in situ carcinoma of the cervix, adequately treated non melanomatous carcinoma of the skin, and other malignancy treated at least 5 years previously with no evidence of recurrence
5. Pre-existing motor/sensory peripheral neuropathy of CTCAE version 3.0 grade >1
6. Patients having received > 3 regimens of chemotherapy
7. Prior therapy with capecitabine and/or vinca-alkaloids
8. History of severe hypersensitivity to vinca alkaloids and/or to fluoropyrimidine or any contra indication to any of the study drugs
9. Known or suspected DPD
10. Pregnant or lactating; With positive pregnancy test at inclusion
11. Female of childbearing potential who is unwilling or unable to use a medically accepted method to avoid pregnancy during the 2 months preceding the start of study treatment, throughout the study period and at least 3 months following the last dose of study treatment
12. Known history of HIV infection
13. Inability to take and/or absorb oral medication
14. Any serious, concurrent uncontrolled medical disorder especially uncontrolled hypercalcaemia, congestive heart failure, uncontrolled high-risk hypertension, arrhythmia, angina pectoris or previous history of myocardial infarction within 6 months prior to randomisation.
15. Prior BMT or autologous stem cell infusion following high-dose chemotherapy.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binghe XU, MD, Study Chair — Cancer Institute & Hospital. Chinese Academy of Medical Sciences, Beijing
Locations (18):
- China (13):
  - Beijing
  - Changchun
  - Chengdu
  - Dalian
  - Fuzhou
  - Hangzhou
  - Harbin
  - Jinan
  - Nanjing
  - Shanghai
  - Shenyang
  - Tianjin
  - Wuhan
- Singapore (2):
  - NUH, Singapore
  - Gleneagles Hospital, Singapore
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A : iv Vinflunine Plus Capecitabine: Vinflunine dose 280 mg/m² on day 1 of each cycle every 3 weeks, Capecitabine 825 mg/m² twice daily orally for 14 consecutive days beginning on day 1 of each cycle followed by 1 week of rest.
  vinflunine: intraveinous administration day 1 once every 3 weeks, 280 mg/m²
  Capecitabine: Arm A : 1650 mg/m² Arm B : 2500 mg/m²
- Arm B : Capecitabine: 1250 mg/m² twice daily orally for 14 consecutive days beginning on day 1 of each cycle followed by 1 week of rest
  Capecitabine: Arm A : 1650 mg/m² Arm B : 2500 mg/m²
Period: Overall Study
Arm/Group | Arm A : iv Vinflunine Plus Capecitabine | Arm B : Capecitabine
Started | 56 | 56
Completed | 0 | 1
Not Completed | 56 | 55
Not completed — Not treated | 0 | 1
Not completed — Progressive disease | 35 | 45
Not completed — Related Adverse events | 7 | 2
Not completed — Non-related adverse events | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 14 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A : iv Vinflunine Plus Capecitabine | Arm B : Capecitabine | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 54 | 109
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Singapore | 4 | 5 | 9
  China | 49 | 46 | 95
  Taiwan | 3 | 5 | 8
Menopausal status [Count of Participants; unit: Participants]
  Menopausal | 31 | 29 | 60
  Non-Menopausal | 25 | 27 | 52
Tumour site - primary cancer [Count of Participants; unit: Participants]
  Right Breast | 23 | 32 | 55
  Left Breast | 33 | 24 | 57

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The primary endpoint for the trial is progression-free survival calculated from the date of randomisation until the date of progression or the date of death whatever the cause of death. Patient who does not progressed will be censored at the date of last tumour assessment or the date of last contact of a follow-up showing no progression.
Time Frame: progression date will be assessed evey 6 weeks starting from the randomization date until first documented progression or date of death from any cause whichever came first assessed up to 3 years
Population: The ITT population, comprised of all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A : iv Vinflunine Plus Capecitabine | Arm B : Capecitabine
Number analyzed (Participants) | 56 | 56
Participants
  Number of events (Participants) | 42 | 46
  Number of censored observations (Participants) | 14 | 10

ADVERSE EVENTS:
Time Frame: 3 years 3 months
Arm/Group | Arm A : iv Vinflunine Plus Capecitabine | Arm B : Capecitabine
All-Cause Mortality (participants affected / at risk) | 26/56 | 32/55
Serious Adverse Events (participants affected / at risk) | 15/56 | 7/55
Other Adverse Events (participants affected / at risk) | 54/56 | 46/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A : iv Vinflunine Plus Capecitabine (N=56) | Arm B : Capecitabine (N=55)
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
ALAT increased (Investigations) | 0 | 1
ASAT increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A : iv Vinflunine Plus Capecitabine (N=56) | Arm B : Capecitabine (N=55)
Nausea (Gastrointestinal disorders) | 13 | 12
Constipation (Gastrointestinal disorders) | 19 | 3
Abdominal pain (Gastrointestinal disorders) | 13 | 3
Vomiting (Gastrointestinal disorders) | 11 | 4
Stomatitis (Gastrointestinal disorders) | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 1
Abdominal distension (Gastrointestinal disorders) | 7 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 2
Gastroesophagal reflux disease (Gastrointestinal disorders) | 3 | 3
Oral pain (Gastrointestinal disorders) | 3 | 0
Weight decreased (Investigations) | 14 | 9
Weight increased (Investigations) | 4 | 13
Neutrophil count decreased (Investigations) | 6 | 0
White blodd cell count decreased (Investigations) | 3 | 1
Fatigue (General disorders) | 14 | 9
Pain (General disorders) | 10 | 1
Oedema pheripheral (General disorders) | 1 | 5
Neuropenia (Blood and lymphatic system disorders) | 11 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Headache (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 4 | 1
Hypoaesthenia (Nervous system disorders) | 1 | 4
Palmer-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 5 | 17
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Oesopharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Early termination of the study. Efficacy analyses were reduced to a descriptive summary of the primary efficacy variable (PFS) in the ITT population. This did not demonstrate any additional benefit of supplementing CAPE with VFL.

Abbreviated CSR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT01953003/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT01953003/SAP_001.pdf